CLINICAL TRIAL: NCT05305040
Title: Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of ALVR105 Posoleucel (ALVR105,Viralym-M) Compared to Placebo for the Prevention of AdV, BKV, CMV, EBV, HHV-6, and JCV Infection and/or Disease, in High-Risk Patients After Allogeneic Hematopoietic Cell Transplant
Brief Title: Study of Posoleucel (ALVR105,Viralym-M) for Multi-Virus Prevention in Patients Post-Allogeneic Hematopoietic Cell Transplant
Acronym: Prevent
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study discontinued as DSMB determined it was futile. No safety concerns were noted.
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P-105-202 Phase 3
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Adenovirus Infection; BK Virus Infection; Cytomegalovirus Infections; Epstein-Barr Virus Infections; Human Herpes Virus-6 Infection; JC Virus Infection
Keywords: Allogeneic Hematopoietic Cell Transplant; ALVR105; Posoleucel; Viralym-M; Virus-specific T cells (VSTs); Cytotoxic T Lymphocytes (CTLs)
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Posoleucel (ALVR105) (Experimental): Administered as 2-4 milliliter infusion, visually identical to placebo
  Interventions: Biological: Posoleucel (ALVR105)
- Placebo (Placebo Comparator): Administered as 2-4 milliliter infusion, visually identical to Posoleucel (ALVR105)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Posoleucel (ALVR105) — Administered as 2-4 milliliter infusion, visually identical to placebo
  Other Names: Viralym-M
  Arms: Posoleucel (ALVR105)
Biological: Placebo — Administered as 2-4 milliliter infusion, visually identical to Posoleucel (ALVR105)
  Arms: Placebo

SUMMARY:
This is a Phase 3 study to evaluate posoleucel (ALVR105, Viralym-M); an allogeneic, off-the-shelf multi-virus specific T cell therapy that targets six viral pathogens: BK virus, cytomegalovirus, adenovirus, Epstein-Barr virus, human herpesvirus 6 and JC virus.

DETAILED DESCRIPTION:
This is a Phase 2/3, multicenter, randomized, double-blind, placebo controlled trial comparing posoleucel to placebo for the prevention of infection or disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV in high-risk adult and pediatric patients after allogeneic HCT.

There are 2 parts to the study, a Phase 3 randomized study cohort described in this posting, and an open label Phase 2 cohort described in NCT04693637, which has completed enrollment. In this Phase 3 part, approximately 302 eligible allogeneic HCT recipients will be enrolled and will receive 7 doses of posoleucel or placebo over 12 weeks, followed by a 12 week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Any age at the day of screening visit.
* No known or suspected clinically significant disease from AdV, BKV, CMV, EBV, HHV-6, and/or JCV
* Within 25 days of receiving a first allogeneic HCT and have demonstrated clinical engraftment at time of dosing
* Meet one or more of the following criteria at the time of randomization:

  * Related (sibling) donor with at least one mismatch at one of these HLA-gene loci: HLA-A, -B or -DR
  * Haploidentical donor
  * Matched or Mismatched unrelated donor
  * Use of umbilical cord blood as stem cell source
  * Ex vivo graft manipulation resulting in T cell depletion
  * Received anti-thymocyte globulin or alemtuzumab (Campath-1H)

Key Exclusion Criteria:

* History of AdV, BKV, CMV, EBV, HHV-6, and/or JCV end-organ disease within 6 months prior to randomization
* Evidence of active Grade >2 acute GVHD
* Presence of non-minor uncontrolled or progressive bacterial, viral or fungal infections
* Known history or current (suspected) diagnosis of Grade ≥3 CRS requiring treatment associated with the administration of peptides, proteins, and/or antibodies
* Ongoing therapy with high-dose systemic corticosteroids (ie, prednisone equivalent dose >1.0 mg/kg/day) within 24 hours prior to dosing
* Relapse of primary malignancy other than minimal residual disease

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (88):
- United States (35):
  - University of Alabama at Birmingham Children's of Alabama, Birmingham, Alabama
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco - Benioff Children's Hospital, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Childrens National Health System, Washington D.C., District of Columbia
  - University of Florida (UF) - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Hospital Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Hospital Cancer Center, Stony Brook, New York
  - Carolinas Medical Center/Levine, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah/Primary Childrens Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Austin Health, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Royal Melbourne Hospital, Parkville
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Belgium (3):
  - A.Z. Sint-Jan Brugge Oostende AV, Bruges
  - Institut Jules Bordet and the Childrens Hospital, Brussels
  - University Hospital Gasthuisberg and Leuven, Leuven
- Canada (6):
  - Alberta Children's Hospital, Calgary
  - Cellular Therapy Program - CHU Sainte-Justine (McGill), Montreal
  - Hopital Maisonneve Rosemont, Montreal
  - The Hospital for Sick Children Blood & Marrow Transplant / Cellular Therapy Program, Toronto
  - UHN Blood and Marrow Transplant (BMT) Program (Princess Margaret) Cancer Center, Toronto
  - Leukemia/ BMT Program of British Columbia - Vancouver General Hospital, Vancouver
- France (7):
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - CHU de Nantes, Nantes
  - AP-HP Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Universitaire Robert Debre, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - IUCT-Oncopole, Toulouse
- Italy (7):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - IRCSS Ospedale Pediatrico Bambino Gesu, Roma
  - University of Sacred Heart Policlinico A. Gemelli, Rome
  - Humanitas Cancer Center, Rozzano
  - Azienda Ospedaliera Universitaria Integrata Verona (AOUI), Verona
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Hwasun
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (4):
  - Institut Catala d'Oncologia, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (9):
  - Acibadem Adana Hospital, Adana
  - Baskent Adana Hospital, Adana
  - Ankara Onkoloji Egitim Ve Arastirma Hastanesi, Ankara
  - Ankara University Hospital, Ankara
  - Gazi University Medical Faculty Hospital, Ankara
  - Medical Park Hospital, Antalya
  - Ege University Medical Faculty, Izmir
  - Anadolu Medical Center Hospital, Kocaeli
  - Inonu University Turgut Özal Medical Centre, Malatya
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol
  - University Hospitals Bristol - Bristol Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Queen Elizabeth University Hospital - Glasgow, Glasgow
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posoleucel (ALVR105), an Off-the-Shelf, Multivirus-Specific T-Cell Therapy, for the Prevention of Viral Infections Post-HCT: Results from an Open-Label Cohort of a Phase 2 Trial Sanjeet S Dadwal, Michael Shuster, Gary Douglas Myers, Keith Boundy, Marshelle Warren, Elizabeth Stoner, Thuy Truong, Joshua A. Hill Blood (2021) 138 (Supplement 1): 1760.
- [Background] Tzannou I, Papadopoulou A, Naik S, Leung K, Martinez CA, Ramos CA, Carrum G, Sasa G, Lulla P, Watanabe A, Kuvalekar M, Gee AP, Wu MF, Liu H, Grilley BJ, Krance RA, Gottschalk S, Brenner MK, Rooney CM, Heslop HE, Leen AM, Omer B. Off-the-Shelf Virus-Specific T Cells to Treat BK Virus, Human Herpesvirus 6, Cytomegalovirus, Epstein-Barr Virus, and Adenovirus Infections After Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2017 Nov 1;35(31):3547-3557. doi: 10.1200/JCO.2017.73.0655. Epub 2017 Aug 7. PMID 28783452
- [Derived] Vasileiou S, Kuvalekar M, Velazquez Y, Watanabe A, Leen AM, Gilmore SA. Phenotypic and functional characterization of posoleucel, a multivirus-specific T cell therapy for the treatment and prevention of viral infections in immunocompromised patients. Cytotherapy. 2024 Aug;26(8):869-877. doi: 10.1016/j.jcyt.2024.03.012. Epub 2024 Mar 19. PMID 38597860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at high risk for viral infection after allogeneic Hematopoietic Cell Transplant were enrolled in the Phase 3 portion of study P-105-202 between Mar 2022 and Jan 2024. The Phase 3 study was discontinued in Dec 2023 after futility analysis of the Primary Outcome Measure. No safety concerns were identified. The Phase 2 portion of study P-105-202 is reported under NCT number NCT04693637.
Pre-assignment Details: A total of 451 participants were enrolled in this Phase 3 study. Due to the early termination of this study, 74 were not dosed. The 377 randomized participants that were dosed comprise the Safety Population.
Groups:
- Posoleucel (ALVR105): Participants received posoleucel administered as 2-4 mL intravenous (IV) infusion once every 14 days for 7 doses.
- Placebo: Participants received placebo administered as 2-4 mL IV infusion once every 14 days for 7 doses.
Period: Overall Study
Arm/Group | Posoleucel (ALVR105) | Placebo
Started (Participants Randomized) | 225 | 226
Participants Dosed (Safety Population) | 188 | 189
Completed | 100 | 101
Not Completed | 125 | 125
Not completed — Not Dosed | 37 | 37
Not completed — Study Closure | 34 | 46
Not completed — Death | 14 | 13
Not completed — Withdrawal by Subject | 15 | 10
Not completed — Other | 13 | 10
Not completed — Primary Malignancy Relapse | 3 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Graft versus host disease | 2 | 0
Not completed — Investigator's Decision | 1 | 1
Not completed — COVID-19 Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: included all participants who received at least one dose of posoleucel or placebo.
Groups:
- Posoleucel (ALVR105): Participants received posoleucel administered as 2-4 mL IV infusion once every 14 days for 7 doses.
- Total: Total of all reporting groups
Arm/Group | Posoleucel (ALVR105) | Placebo | Total
Number analyzed (Participants) | 188 | 189 | 377
Age, Continuous [Median (Full Range); unit: years] | 55.0 [1 to 77] | 53.0 [0 to 75] | 54.0 [0 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 66 | 144
  Male | 110 | 123 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 24 | 37
  Not Hispanic or Latino | 143 | 144 | 287
  Unknown or Not Reported | 32 | 21 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 1 | 2
  Asian | 25 | 21 | 46
  Black or African American | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 118 | 131 | 249
  Other | 9 | 8 | 17
  Unknown | 27 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Clinically Significant Infections or Episodes of End-Organ Disease Through Week 14
Description: The average number of clinically significant infections or episodes of end-organ disease per participant due to Adenovirus (AdV), BK virus (BKV), Cytomegalovirus (CMV), Epstein-Barr virus (EBV), Human herpes virus 6 (HHV-6), or JC virus (JCV).
Time Frame: Through Week 14
Population: Includes modified Intent-to-Treat (mITT) Population comprised of all randomized participants who received study drug and completed through Week 14 visit.
Measure: Mean (Standard Deviation); unit: Infections/Episodes per participant
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 159 | 155
Infections/Episodes per participant | 0.2 (0.44) | 0.2 (0.42)
Statistical Analysis 1: Comparison: Posoleucel (ALVR105) vs Placebo; Test type: Superiority; p = 0.5603, ANCOVA — 1-sided p-value; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.09 to 0.10], Standard Error of Mean 0.049

2. Secondary Outcome: Average Number of Clinically Significant Infections or Episodes of End-Organ Disease Through Week 26
Description: The number of clinically significant infections or episodes of end-organ disease per participant due to AdV, BKV, CMV, EBV, HHV-6, or JCV.
Time Frame: Through Week 26
Population: Data not collected due to early termination after DSMB futility analysis concluded the study was unlikely to meet its primary endpoint.
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Clinically Significant Infections or Episodes of End-Organ Disease Due to Each Virus
Description: The number of participants with clinically significant infections or episodes of end-organ disease due to each of the following viruses: AdV, BKV, CMV, EBV, HHV-6, or JCV.
Time Frame: Through Week 14
Population: Includes mITT Population comprised of all randomized participants who received study drug and completed through Week 14 visit.
Measure: Number; unit: participants
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 159 | 155
participants
  AdV | 3 | 2
  BKV | 2 | 2
  CMV | 16 | 19
  EBV | 10 | 6
  HHV-6 | 0 | 0
  JCV | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Week 26.
Description: Adverse events are reported for the Safety Population which included all participants who received at least one dose of posoleucel or placebo.
Groups:
- Placebo: Participants received placebo administered as a 2-4 mL IV infusion once every 14 days for 7 doses.
Arm/Group | Posoleucel (ALVR105) | Placebo
All-Cause Mortality (participants affected / at risk) | 18/188 | 19/189
Serious Adverse Events (participants affected / at risk) | 88/188 | 86/189
Other Adverse Events (participants affected / at risk) | 180/188 | 184/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=188) | Placebo (N=189)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Warm autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Strabismus (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 12
Disease progression (General disorders) | 3 | 0
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 7 | 7
Acute graft versus host disease in skin (Immune system disorders) | 4 | 2
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 3
Graft versus host disease in liver (Immune system disorders) | 2 | 2
Acute graft versus host disease (Immune system disorders) | 1 | 2
Graft versus host disease (Immune system disorders) | 1 | 2
Graft versus host disease in skin (Immune system disorders) | 1 | 2
Acute graft versus host disease in liver (Immune system disorders) | 2 | 0
Chronic graft versus host disease in skin (Immune system disorders) | 0 | 2
Autoimmune disorder (Immune system disorders) | 0 | 1
Chronic graft versus host disease (Immune system disorders) | 0 | 1
Chronic graft versus host disease in liver (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 5 | 4
Pneumonia (Infections and infestations) | 4 | 4
Cytomegalovirus infection (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 5 | 2
Bacteraemia (Infections and infestations) | 2 | 4
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 4
Adenovirus infection (Infections and infestations) | 1 | 3
Epstein-Barr viraemia (Infections and infestations) | 2 | 2
Cytomegalovirus viraemia (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2
Device related bacteraemia (Infections and infestations) | 0 | 2
Epstein-Barr virus infection reactivation (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Norovirus infection (Infections and infestations) | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 2
Toxoplasmosis (Infections and infestations) | 0 | 2
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 1
Adenoviral haemorrhagic cystitis (Infections and infestations) | 0 | 1
Adenovirus reactivation (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Clostridial sepsis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Human bocavirus infection (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection reactivation (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Enterobacter test positive (Investigations) | 1 | 0
Epstein-Barr virus antigen positive (Investigations) | 1 | 0
Epstein-Barr virus test positive (Investigations) | 0 | 1
Herpes simplex test positive (Investigations) | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Precursor T-lymphoblastic lymphoma/leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebellar haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Transient aphasia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Cardio-respiratory arrest with sepsis (Cardiac disorders) | 0 | 1
Fever and rigors (General disorders) | 1 | 0
Hospitalization for nausea and vomiting (Gastrointestinal disorders) | 0 | 1
Positive cultures from indwelling CVAD (General disorders) | 0 | 1
Sepsis with multiple organ failure (Infections and infestations) | 1 | 0
Sepsis with fever and rigor (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=188) | Placebo (N=189)
Anaemia (Blood and lymphatic system disorders) | 26 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 9
Neutropenia (Blood and lymphatic system disorders) | 12 | 7
Dry eye (Eye disorders) | 5 | 13
Diarrhoea (Gastrointestinal disorders) | 46 | 37
Nausea (Gastrointestinal disorders) | 36 | 22
Vomiting (Gastrointestinal disorders) | 29 | 21
Abdominal pain (Gastrointestinal disorders) | 25 | 16
Constipation (Gastrointestinal disorders) | 12 | 10
Pyrexia (General disorders) | 33 | 36
Fatigue (General disorders) | 22 | 17
Oedema peripheral (General disorders) | 17 | 20
Asthenia (General disorders) | 11 | 8
Acute graft versus host disease in skin (Immune system disorders) | 36 | 27
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 24 | 16
Graft versus host disease in skin (Immune system disorders) | 15 | 15
Acute graft versus host disease (Immune system disorders) | 11 | 7
Hypogammaglobulinaemia (Immune system disorders) | 6 | 12
Cytomegalovirus infection (Infections and infestations) | 13 | 18
Pneumonia (Infections and infestations) | 11 | 14
COVID-19 (Infections and infestations) | 13 | 11
Cytomegalovirus infection reactivation (Infections and infestations) | 10 | 11
Upper respiratory tract infection (Infections and infestations) | 5 | 14
Sepsis (Infections and infestations) | 10 | 3
Fall (Injury, poisoning and procedural complications) | 8 | 10
Blood creatinine increased (Investigations) | 30 | 22
Platelet count decreased (Investigations) | 22 | 15
Alanine aminotransferase increased (Investigations) | 14 | 16
Aspartate aminotransferase increased (Investigations) | 9 | 11
White blood cell count decreased (Investigations) | 12 | 8
Neutrophil count decreased (Investigations) | 10 | 8
Decreased appetite (Metabolism and nutrition disorders) | 18 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11
Headache (Nervous system disorders) | 22 | 22
Tremor (Nervous system disorders) | 14 | 11
Dizziness (Nervous system disorders) | 10 | 12
Insomnia (Psychiatric disorders) | 11 | 7
Acute kidney injury (Renal and urinary disorders) | 14 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 14
Rash (Skin and subcutaneous tissue disorders) | 16 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 12
Erythema (Skin and subcutaneous tissue disorders) | 11 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 9
Hypertension (Vascular disorders) | 16 | 7

LIMITATIONS AND CAVEATS:
The Sponsor decided to discontinue the Phase 3 part of the trial on 22 Dec 2023 following a pre-planned DSMB futility analysis concluding the study was unlikely to meet its primary endpoint; no safety concerns were identified. Data was not collected for efficacy analyses at Week 26 as planned. Participants were monitored through Week 26 for safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT05305040/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT05305040/SAP_001.pdf